CLINICAL TRIAL: NCT05420922
Title: Efficacy and Safety of Immune Checkpoint Inhibitors (ICIs) and Tyrosine Kinase Inhibitors (TKIs) Therapy for Hepatocellular Carcinoma (HCC)：a Multicenter, Retrospective Study on the Real-world in China
Brief Title: Real-world Study of Efficacy and Safety of ICIs and TKIs Therapy for HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Professor, Tongji Hospital
Other Study IDs: CHL2022
Record Dates: First submitted 2022-05-26; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma; Programmed Cell Death 1; Effects of Immunotherapy
Keywords: Lenvatinib; Sorafenib; Programmed Cell Death 1; Real-world study; transcatheter arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Systemic therapy: ICIs (PD1 or PDL-1)+TKIs (Lenvatinib or Sorafenib)
  Interventions: Drug: Lenvatinib Oral Product; Drug: PD-1 inhibitor
- Local treatment: local treatment include: TACE, HAIC, RF Ablation, Microwave Ablation, Radiotherapy, etc.
  Interventions: Procedure: Local treatment
- Triple therapy: Systemic therapy plus Local treatment:
  ICIs (PD1 or PDL-1)+TKIs (Lenvatinib or Sorafenib) plus local treatment (TACE, HAIC, RF Ablation, Microwave Ablation, Radiotherapy, etc)
  Interventions: Drug: Lenvatinib Oral Product; Drug: PD-1 inhibitor; Procedure: Local treatment

INTERVENTIONS:
Drug: Lenvatinib Oral Product — Lenvatinib or Sorafenib
  Groups: Systemic therapy; Triple therapy
Drug: PD-1 inhibitor — Programmed cell death protein-1 (PD-1) or Programmed cell death ligand 1 (PDL-1
  Groups: Systemic therapy; Triple therapy
Procedure: Local treatment — Local treatment include: TACE, HAIC, RF Ablation, Microwave Ablation, Radiotherapy, etc.
  Groups: Local treatment; Triple therapy

SUMMARY:
China is a high-risk area of Hepatocellular Carcinoma (HCC). Although Chinese population accounts for 18.4% of the global population, the number of new HCC patients accounting for about half of the global, which seriously threatens the lives and health of the people. The investigators establish multi-center, retrospective research methods, collecting the data of HCC treatment with system treatment (ICIs and TKIs) plus or without local treatment in the last 3 years, comprehensive assessment of their efficacy and safety, explore whether the efficacy of system treatment combination local treatment showed better effect compared with system or local monotherapy. Our study will find a new way to improve the prognosis of HCC patients.

DETAILED DESCRIPTION:
This was a multi-center, retrospective study involving 2000 patients with HCC receiving ICIs (Programmed cell death protein-1 (PD-1) or Programmed cell death ligand 1 (PDL-1)) and TKIs (Lenvatinib or Sorafenib), ICIs and TKIs plus local treatment (TAC, Hepatic artery infusion chemotherapy (HAIC), radiofrequency (RF) ablation, microwave ablation, radiotherapy, etc.), and local monotherapy between Jan, 2019 and Dec, 2021 in China. Efficacy was evaluated with objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), time to tumor progression (TTP), and 1year and 2 years overall survival (OS). Treatment-related adverse events (TRAEs) were recorded and graded. Efficacy and safety of three groups were compared. Stratified analysis was performed according to patients baseline characteristics and medication regimen for combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatocellular carcinoma
* Treated with ICIs (PD-1 or PDL-1) therapy plus TKIs (Lenvatinib or sorafenib)
* Treated with local therapy (TACE, HAIC, RF ablation, microwave ablation, radiotherapy, etc)
* Treated Treated with ICIs plus TKIs and local therapy
* Have complete medical record that can complete the OR or 1 year OS assessment and follow-up.

Exclusion Criteria:

* Patients who do not have complete medical record and follow-up information after treatment；
* The researchers have evidence that it is not suitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma patients using ICIs (PD-1 or PDL-1) therapy plus TKIs (Lenvatinib or sorafenib), ICIs plus TKIs with local therapy (TACE, HAIC, RF ablation, microwave ablation, etc), local therapy only
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The objective response rate (ORR) | 8 weeks
  ORR in three groups were compared
The overall survival (OS) | 12 months
  1 year OS in three groups were compared
The treatment-related adverse events (TRAEs) | 12 months
  Rate of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
The progression-free survival (PFS) | 8 weeks
  ORR in three groups were compared

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided whether it needs to cooperate with other PI.